CLINICAL TRIAL: NCT07361978
Title: The Effect of Purse-Lip Breathing Exercise on Anxiety and Physiological Parameters Post-Bronchoscopy in Patients With COPD: A Randomized Controlled Trial
Brief Title: The Effect of Pursed-Lip Breathing Exercise on Anxiety and Physiological Parameters Post-Bronchoscopy in Patients With COPD: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Ruhat Tilki, Research Assistant, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 133.2025fbu
Record Dates: First submitted 2025-12-31; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: COPD
Keywords: copd; pursed-lip breathing; Nursing care; anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (No Intervention): There will be normal nursing care
- PLB + Routine Care (Experimental): Following a conscious inhalation through the nose, it involves exhaling slowly and in a controlled manner through pursed lips; this prolongs the exhalation phase compared to the normal inspiration-exhalation ratio.
  Interventions: Other: Pursed-Lip Breathing exercise and Routine Care

INTERVENTIONS:
Other: Pursed-Lip Breathing exercise and Routine Care — Pursed-Lip Breathing exercise will be done. Following a conscious inhalation through the nose, it involves exhaling slowly and in a controlled manner through pursed lips; this prolongs the exhalation phase compared to the normal inspiration-exhalation ratio.
  Arms: PLB + Routine Care

SUMMARY:
This randomized controlled trial investigates the effect of Pursed Lip Breathing (PLB) on anxiety levels and physiological parameters in patients with Chronic Obstructive Pulmonary Disease (COPD) following bronchoscopy. While PLB is known to improve oxygenation and ventilation in pulmonary rehabilitation, its specific impact on the immediate recovery period after bronchoscopy is understudied. The study aims to determine if nurse-led PLB intervention significantly improves heart rate, blood pressure, oxygen saturation, and reduces anxiety compared to standard care.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD), which ranks among the leading causes of morbidity and mortality worldwide, is expected to have increasingly negative consequences. There are over 600 million COPD patients worldwide and approximately 2-3 million in Turkey. COPD requires a complex and long-term response that coordinates the contributions of a wide range of professionals, specific types of medication, and appropriate monitoring equipment, and this care should ideally be integrated into a system that promotes patient empowerment. The associated treatment process involves repeated hospital admissions, which impose high economic costs on countries.

In the dynamic environment of critical care medicine, bedside bronchoscopy has emerged as a crucial diagnostic and therapeutic tool that bridges the gap between traditional pulmonary interventions and the urgent needs of critically ill patients. Bronchoscopy allows direct visualization of the airways and lung parenchyma and can be useful in evaluating various bronchopulmonary conditions and diseases, including foreign bodies, tumors, infectious and inflammatory processes, airway obstruction, and bronchopulmonary hemorrhage. Bronchoscopy may also be associated with other complications and discomforts beyond existing respiratory system problems.

Teaching patients breathing exercises is another nursing intervention that can increase oxygenation and reduce dyspnea. Various breathing exercises are available, including PLB. PLB is a breathing technique used to improve oxygenation and ventilation. This breathing technique involves consciously inhaling through the nose, followed by a slow and controlled exhalation through pursed or pinched lips, which prolongs the exhalation phase compared to the normal inspiration-exhalation ratio.

Nurses' ability to promptly recognize distress enables intervention teams to respond quickly and prevent further deterioration. The literature shows that pursed-lip breathing improves vital signs and oxygenation in COPD rehabilitation and during the recovery process after bronchoscopy. In a recent study, patients who practiced pursed-lip breathing during the post-bronchoscopy period showed significant improvements in parameters such as oxygen saturation, pulse rate, and blood pressure compared to the control group. However, studies examining the effect of this technique on anxiety and immediate physiological parameters in COPD patients during the bronchoscopy procedure are limited. This study was designed as a randomized controlled trial to determine the effect of PLB application on anxiety levels and physiological parameters (heart rate, blood pressure, oxygen saturation) in patients with COPD after bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD
* Patients undergoing elective bronchoscopy under sedation
* Patients aged 18 - 80 years
* Patients who are fully oriented, conscious, and able to communicate

Exclusion Criteria:

* Patients undergoing emergency bronchoscopy
* Patients with hemodynamic instability prior to the procedure (systolic blood pressure <90 mmHg or >180 mmHg)
* Patients with severe hearing or cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in State Anxiety Level | Baseline (Pre-procedure) and immediately after the bronchoscopy procedure (up to 30 minutes).
  Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI), specifically the State Anxiety subscale (STAI-S). The scale consists of 20 items. Total scores range from a minimum of 20 to a maximum of 80. Higher scores indicate higher levels of anxiety (worse outcome), while lower scores indicate lower levels of anxiety.

SECONDARY OUTCOMES:
Change in Oxygen Saturation (SpO2) | Baseline, during the procedure, and immediately after the procedure. Baseline, during the procedure, and immediately after the procedure. (30 minutes before and after the procedure.)
  Measured via pulse oximetry. Values are recorded as a percentage (%). Higher values indicate better physiological oxygenation status. Unit of measure: Percentage of oxygen saturation
Change in Heart Rate | Baseline, during the procedure, and immediately after the procedure (up to 30 minutes).
  Measured via pulse oximetry or cardiac monitor. Values are recorded as beats per minute (bpm). Lower values (within normal range) generally indicate lower physiological stress.
Change in Systolic Blood Pressure | Baseline (pre-procedure), during the procedure, and immediately after the procedure (up to 30 minutes).
  Measured via non-invasive blood pressure cuff. Values are recorded in millimeters of mercury (mmHg).
Change in Diastolic Blood Pressure | Baseline (pre-procedure), during the procedure, and immediately after the procedure (up to 30 minutes).
  Measured via non-invasive blood pressure cuff. Values are recorded in millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Süreyyapaşa Göğüs Hastalıkları ve Göğüs Cerrahisi EAH, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No